CLINICAL TRIAL: NCT07103681
Title: Observational Study to Investigate the Effect of White Matter Tract Distortion and Neurodegenerative Biomarkers on Shunt-responsiveness in Idiopathic Normal Pressure Hydrocephalus (iNPH)
Brief Title: White Matter Distortion and Dementia Biomarkers in Normal Pressure Hydrocephalus (NPH)
Acronym: OWN-NPH
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Michael J. Fox Foundation for Parkinson's Research (Other); University College, London (Other); University of Edinburgh (Other); King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 311620; W0300981 (Other Grant/Funding Number: Medical Research Council (MRC))
Record Dates: First submitted 2025-03-03; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: hydrocephalus; activity monitors; gait impairment; shunt surgery; protokinetic; normal pressure hydrocephalus; shunt-responsiveness; white matter tractography; diffusion tensor imaging; neurodegenerative; NPH
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus | interventions — Ventriculoperitoneal Shunt

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, CSF, brain and skin will be retained for 10 years following the study end and keeping with the ICL policies. Unless used in other ongoing studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group 1: Group 1 includes adults over 60 years old diagnosed with late-onset communicating hydrocephalus, characterised by gait apraxia, with or without cognitive impairment and urinary dysfunction. Eligibility is confirmed through clinical imaging showing an Evan's index >0.3 and an iNPH Radscale score >4. Individuals with recent severe head trauma, high-pressure hydrocephalus, or alternative causes for similar symptoms are excluded. This criteria for group 1 ensures a distinct group for studying the late-onset, communicating form of the condition.
  Interventions: Procedure: Ventriculoperitoneal Shunt (VP); Procedure: Brain and Skin Biopsy; Diagnostic Test: MRI Brain
- Group 2: Group 2 will include 30 adult patients with asymptomatic chronic hydrocephalus, non-hydrocephalus dementia and healthy controls.

INTERVENTIONS:
Procedure: Ventriculoperitoneal Shunt (VP) — VP Shunt surgery involves surgical insertion of a catheter (tube) to divert brain fluid from the cerebral ventricles to the abdominal peritoneum. This will be performed in Group 1 patients as clinically indicated.
  Other Names: VP Shunt
  Groups: Group 1
Procedure: Brain and Skin Biopsy — Brain and skin biopsy's may be taken during the VP shunt to assist in histological analysis for neurodegenerative changes.
  Groups: Group 1
Diagnostic Test: MRI Brain — MRI brain with diffusion imagining will be performed before and after shunt surgery.
  Groups: Group 1

SUMMARY:
Idiopathic Normal Pressure Hydrocephalus (iNPH) is a progressive condition of the elderly that results in severe disability. iNPH can dramatically respond to Cerebral spinal fluid(CSF)-shunting where excess ventricular fluid is diverted from the brain. Not all patients with iNPH respond to CSF-shunting however. The reasons for this are uncertain.

Aim 1: To understand if specific nerve pathways (white matter tracts) that are near ventricles are damaged in patients that respond to shunting as opposed to those that do not.

Aim 2: Can we explain shunt non-responsiveness by screening for dementia like illnesses (neurodegeneration) using a large array of methods.

Aim 3: To understand whether wearable activity and bed sleep monitors are palatable in a NPH population and to understand if these metrics relate to quality of life.

Aim 4: To see whether self-administered digital cognitive assessments can measure improvements pre and post surgery.

DETAILED DESCRIPTION:
This single-centre observational cohort study will follow 50 patients diagnosed with symptomatic Normal Pressure Hydrocephalus (NPH) (idiopathic or late presenting congenital hydrocephalus and not secondary hydrocephalus) through their clinical journey, from initial assessment to post-CSF shunt surgery or a time when surgery is decided against. Separate groups of 50 asymptomatic individuals with chronic hydrocephalus and non-hydrocephalus individuals will act as controls.

Participants will undergo comprehensive clinical assessments including gait, cognitive and urinary evaluations, quality of life measures, serum and CSF degenerative biomarker analysis, diffusion-weighted Magnetic Resonance Imaging (MRI) and optional brain and skin biopsies. Data collection will focus on capturing changes in clinical presentation and imaging findings before and after shunting. REDCap will be utilised as the primary tool for data storage.

Primary outcome measures assess pre and post-shunting imaging changes in shunt-responders and non-responders. Shunt response will be defined as 10% improvement in gait speed. Secondary outcomes evaluate the relationship between biomarkers and clinical outcomes. Longitudinal data will help identify factors distinguishing responders from non-responders, with descriptive and inferential statistics used.

ELIGIBILITY:
Group 1 (communicating hydrocephalus):

Inclusion Criteria:

* Adult patients >60
* With gait apraxia
* With or without cognitive impairment
* Urinary dysfunction
* Communicating Hydrocephalus

Exclusion Criteria:

* Asymptomatic hydrocephalus
* High pressure-hydrocephalus
* Serious head injury within 5 years of presentation or a clear secondary cause (e.g. brain infection)
* History of childhood gait disturbance
* Clear alternative explanation for symptoms (e.g. Parkinson's disease with limb rigidity, peripheral neuropathy with sensory ataxia, cervical myelopathy).
* Too frail for shunt surgery
* Medically unstable (e.g. active angina, respiratory disease, recurrent delirium, active epilepsy).
* Unable to tolerate MRI brain imaging
* Unable to have a lumbar puncture
* Immobile
* Unable to attend the hospital for study visits

Group 2 (asymptomatic and non-hydrocepahlus dementia and healthy controls):

Inclusion Criteria (Any of the following):

* Healthy Carers
* Members of the Public
* Staff of Imperial College/ICHT
* Non-NPH Dementias (including Alzheimer's disease or vascular dementia)
* Asymptomatic Hydrocephalus

Exclusion Criteria:

- Unable to attend the hospital for study visits

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hydrocephalus, neurodegenerative disease and healthy controls will be recruited by Dr Chris Carswell at Imperial College Hospital NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
White Matter Pathway Diffusion Metrics | Perioperative
  Change from baseline in diffusion tensor imaging (DTI) metrics of white matter pathways (e.g. FA, AD, RD) before and after shunt surgery. The following tracts will be studied: corpus collosum, internal capsule, corona radiata and anterior thalamic radiation.

SECONDARY OUTCOMES:
Neurodegenerative Biomarkers and CSF-shunt responsiveness | Perioperative
  Composite degenerative index (plasma abeta, GFAP, Ptau217, NfL, CSF synuclein RT QuIC and brain and skin histology) will be generated and compared between CSF shunt-responsive and CSF non-responsive groups.
Serum Neurodegenerative Biomarkers | From enrolment, at periprocedural and up to 27 weeks
  The serum biomarkers will measure a-beta (pg/ml), G-FAB (pg/ml), NfL (pg/ml) and p-tau217 (pg/ml).
Sleep Monitoring | From enrolment and through study completion, an average of 1 year
  The Withings' Sleep mats are devices designed to track sleep patterns. Participants will be offered under mattress sleep monitors capable of showing time spent in bed and analyse sleep cycles.
Activity Monitoring | From enrolment and through study completion, an average of 1 year
  The Withings' Activity Monitors are devices designed to track physical activity and heart rate. Participants will be offered wrist activity monitors which capture data on steps taken, calories burned and overall movement throughout the day, providing insights into daily activity levels.
Tinetti Performance Oriented Mobility Assessment Score (balance) | From enrolment, at periprocedural and up to 27 weeks
  Total scores range from 0 to 16, with higher scores indicating better outcomes of balance performance.
Tinetti Performance Oriented Mobility Assessment Score (Gait) | From enrolment, at periprocedural and up to 27 weeks
  Total scores range from 0 to 12, with higher scores indicating better outcomes of gait performance.
International Consultation on Incontinence Questionnaire for Urinary Incontinence Short Form (ICIQ UI SF) | From enrolment, at periprocedural and up to 27 weeks.
  The assessment measures the frequency and severity of urinary incontinence. The total scores range from 0-21. Higher scores indicate worse bladder symptoms.
International Consultation on Incontinence Questionnaire for Bowels (ICIQ-B) | From enrolment, at periprocedural and up to 27 weeks.
  The assessment measures the pattern and control of bowel incontinence. The total scores for bowel pattern ranges from 1-21 and bowel control ranges from 0-28. Higher scores indicate worse bowel symptoms.
International Consultation of Incontinence Questionnaire for Sexual Function | From enrolment, at periprocedural and up to 27 weeks.
  The assessment measures the severity and bother of sexual function. The scores for sexual function range from 1-5 and are assessed on an individual basis. Higher scores indicate worse sexual function.
International Consultation of Incontinence Questionnaire for Quality of Life | From enrolment, at periprocedural and up to 27 weeks.
  The assessment measures the quality of life bladder, bowels and sexual function has on the individual. The scores suggest how much they bother the participant and it ranges from 0-10. Higher bother scores indicate lower quality of life.
Overactive Bladder Symptoms (OAB) | From enrolment, at periprocedural, and up to 27 weeks.
  The total score ranges from 0 to 15, with higher scores indicating worse bladder severity symptoms.
Kubo scale | From enrolment, at periprocedural and up to 27 weeks.
  Assesses gait disturbance, cognitive impairment and urinary disturbance. Total scores range from 0 to 12, with higher scores indicating better outcomes.
Patient Health Questionnaire-9 (PHQ-9) | From enrolment, at periprocedural and up to 27 weeks.
  Assesses the severity of depression. Total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
Generalised Anxiety Disorder-7 (GAD-7) | From enrolment, at periprocedural and up to 27 weeks.
  Assesses the severity of anxiety symptoms. Total scores range from 0 to 21, with higher scores indicating more severe anxiety.
Sintonen 15D | From enrolment, at periprocedural and up to 27 weeks.
  Overall score adds 15 metrics of quality of life. Total scores range from 75-15 with lower scores indicating better quality of life.
PSP QoL | From enrolment, at periprocedural and up to 27 weeks.
  Overall score adds 45 metrics of quality of life using a Likert scale to score from 0-5. Total scores range from 0-225 with lower scores indicating better quality of life.
Rockwood Clinical Frailty Scale Score | From enrolment, at periprocedural and up to 27 weeks.
  Frailty rating score in older adults. Total scores range from 1 to 9 with higher indicating greater frailty.
Addenbrooke's Cognitive Examination ||| (ACE-|||) | From enrolment, at periprocedural and up to 27 weeks.
  Total score evaluates cognitive functions including memory, language, visuospatial, attention and language. Total scores range from 0 to 100, with higher scores indicating better cognitive function.
Cognitron Cognitive Assessment Platform | From enrolment, at periprocedural and up to 27 weeks.
  Includes a total score of a collection of cognitive tests to assess various cognitive domains in those with NPH pre and post surgery. There are specific domain specific scores.
PKMAS Gait Analysis Software | From enrolment, at periprocedural and up to 27 weeks.
  Objective gait metric data is taken from the Protokinetics gait mat to analyse gait parameters of those with NPH. These metrics include, all aspects of gait (e.g. foot length, gait velocity, stride length)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared with collaborators if it is within the remit of the ethics approval and depending on the nature of the collaboration.